CLINICAL TRIAL: NCT02029950
Title: A Phase I Study of Pomalidomide Given at the Time of Lymphocyte Recovery Following Induction Timed Sequential Chemotherapy With Cytarabine, Daunorubicin and Etoposide (AcDVP16) in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML) and High-Risk MDS
Brief Title: Pomalidomide After Combination Chemotherapy in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02426; NCI-2013-02426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); J13128; NA_00089739; 9524 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 9524 (Other: CTEP); P30CA006973 (NIH); U01CA070095 (NIH); UM1CA186691 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia-2; High Risk Myelodysplastic Syndrome; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myeloproliferative Disorders | interventions — Cytarabine; Daunorubicin; Etoposide; Idarubicin; 4-demethoxydaunorubicin bis(hydrazone); pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (combination chemotherapy, pomalidomide) (Experimental): See Detailed Description
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Etoposide; Drug: Idarubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Pomalidomide

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Idarubicin Hydrochloride — Given IV
  Other Names: Idamycin; Idamycin PFS; Idarubicin HCl; IMI-30; SC-33428; Zavedos
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase I trial studies the side effects and best dose of pomalidomide after combination chemotherapy in treating patients with newly diagnosed acute myeloid leukemia or high-risk myelodysplastic syndrome. Drugs used in chemotherapy, such as cytarabine, daunorubicin hydrochloride, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Pomalidomide may kill cancer cells by stopping blood flow to the cancer and by stimulating white blood cells to kill cancer cells. Giving more than one drug (combination chemotherapy) and pomalidomide may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) of pomalidomide when given at the time of early lymphocyte recovery following intensive induction timed sequential therapy (TST) with cytarabine (cytosine arabinoside), daunorubicin hydrochloride (daunorubicin) and etoposide (AcDVP-16) in patients with newly diagnosed intermediate- and poor-risk acute myeloid leukemia and high-risk myelodysplastic syndrome (MDS).

II. To evaluate the safety, tolerability and toxicity of pomalidomide given at the time of early lymphocyte recovery following induction AcDVP-16 chemotherapy in adults with newly diagnosed intermediate- and poor-risk acute myeloid leukemia and high-risk MDS.

SECONDARY OBJECTIVES:

I. To evaluate the safety, tolerability and toxicity of pomalidomide given as a continuation therapy following induction and/or consolidation chemotherapy in adults with newly diagnosed intermediate- and poor-risk acute myeloid leukemia and high-risk MDS.

II. To document responses (complete remission [CR], CR with incomplete count recovery [CRi], partial remission [PR]) to AcDVP-16 followed by pomalidomide at the time of lymphocyte recovery in newly diagnosed adults with intermediate- and poor-risk acute myeloid leukemia (AML) and high-risk MDS, including duration of response, disease-free and overall survival.

III. Correlative pharmacodynamics studies: a) to characterize the effects of pomalidomide on the functional dynamics of different lymphocyte subpopulations (effector T [Teff], regulatory T [Treg], natural killer [NK] cells) and its impact on tumor-associated antigen (TAA)-specific T cell immunity when given following induction and as a maintenance; b) to examine for the presence of minimal residual disease (MRD) before and after pomalidomide administration during induction and continuation therapy; c) to examine cereblon expression in primary leukemia cells at diagnosis and in sorted T cells prior to and after pomalidomide treatment.

OUTLINE: This is a dose-escalation study of pomalidomide.

INDUCTION: Patients receive cytarabine intravenously (IV) continuously and daunorubicin hydrochloride IV on days 1-3 (patients may otherwise receive idarubicin hydrochloride IV over 10-15 minutes on days 1-3 if daunorubicin hydrochloride is unavailable), and etoposide IV over 3 hours on days 8-10. At the time of early lymphocyte recovery (after day +14), patients also receive pomalidomide orally (PO) for 10-21 days.

CONSOLIDATION: Patients achieving CR or CRi receive cytarabine based treatment at the discretion of the treating investigator, with possible regimens comprising cytarabine IV continuously on days 1-3, and 10-12 and daunorubicin hydrochloride IV on days 1-3, or high- or medium-dose cytarabine IV every 12 hours on days 1, 3, and 5 for 1-4 courses.

CONTINUATION: Patients achieving CR or CRi who did not undergo allogeneic stem cell transplant receive pomalidomide PO daily on days 1-21 beginning 6 weeks following blood count recovery. Treatment repeats every 4-6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed:

  * Pathologically confirmed intermediate or poor risk newly diagnosed AML (subtypes M0, 1, 2, 4-7), but excluding newly diagnosed core-binding factor (CBF) (t(8;21) or M4eo subtype (inv(16) or t(16;16) AMLs and acute promyelocytic leukemia (acute promyelocytic leukemia [APL], M3)
  * MDS with high risk features as defined by intermediate (INT)-2 or high International Prognostic Scoring System (IPSS) score with > 10% blasts in the bone marrow
  * Chronic myelomonocytic leukemia-2 (CMML-2) defined as having > 10% blasts (including promonocytes) in the bone marrow or 5-19% blasts (including promonocytes) in the peripheral blood
* Patients who have received hydroxyurea alone or have received non-cytotoxic therapies previously for treatment of MDS or myeloproliferative neoplasm (MPN) (e.g. azacitidine, decitabine, histone deacetylase inhibitors, tyrosine kinase inhibitors, hematopoietic growth factors, interferon, lenalidomide, thalidomide) will be eligible for this trial as long as immunomodulatory drugs (e.g. lenalidomide, thalidomide) have not been used in the past 3 months
* Patients must be off all non-cytotoxic chemotherapies or biologic agents (e.g. azacitidine, decitabine, histone deacetylase inhibitors, tyrosine kinase inhibitors, hematopoietic growth factors, interferon, but excluding hydroxyurea and cyclophosphamide) for at least 2 weeks prior to starting induction chemotherapy
* Patients must be off radiation therapy or chemotherapy 4 weeks (6 weeks for nitrosoureas or mitomycin C) of starting induction chemotherapy
* All adverse events (excluding alopecia, acne, rash) due to agents administered more than 2 weeks earlier should recover to =< grade 1; patients with hematologic malignancies are expected to have hematologic abnormalities at study entry; these abnormalities which are thought to be primarily related to the underlying leukemia, are not considered to be toxicities (adverse events [AE]) and do not need to resolve to =< grade 1
* Patients with therapy-related AML or MDS should have not received prior cumulative anthracycline (daunorubicin equivalent) lifetime dose > 450 mg/m^2
* Cytoreduction allowed:

  * Hydroxyurea, corticosteroids, leukapheresis can be used prior to start of induction chemotherapy
  * Cyclophosphamide up to dose 50-60 mg/kg is allowed for cytoreduction, but must be given at least 7+/- 2 days before start of induction chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Total bilirubin < 2.0 mg/dL unless due to Gilbert's disease, hemolysis or leukemia
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional upper limit of normal unless due to leukemic infiltration
* Creatinine =< 2.0 mg/dL
* Left ventricular ejection fraction >= 45%
* Female who is able to become pregnant must have a negative pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours of starting pomalidomide; female who is able to become pregnant must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective and one additional effective method at the same time; female who is able to become pregnant must agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with female who is able to become pregnant even if they had vasectomy for the duration of study participation, and 28 days after completion of pomalidomide administration; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure while taking pomalidomide; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

  * A female who is able to become pregnant is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Ability to understand and the willingness to sign a written informed consent document; consent will be obtained by day 14 of AcDVP-16 induction regimen
* Known human immunodeficiency virus (HIV) infected patients (HIV testing will not be performed as a part of screening) on combination antiretroviral therapy are eligible for inclusion; the use of zidovudine is not allowed

Exclusion Criteria:

* Patients who are receiving any other investigational agents or who have received pomalidomide in the past
* Patients with known active central nervous system leukemia should be excluded from this clinical trial; patient receiving intrathecal chemotherapy prophylaxis should not receive pomalidomide for >= 3 days after administration
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pomalidomide (e.g. lenalidomide, thalidomide) or other agents used in study
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide or similar drugs in the past
* Uncontrolled intercurrent illness including, but not limited to, active and uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, mental deficits, psychiatric illness or history or social situations that would limit compliance with study requirements; patients with infection under active treatment and controlled with antibiotics are eligible
* Any other medical condition that in opinion of investigator would place patient at increased risk for toxicity during pomalidomide treatment (i.e. history of recurrent or serious thromboembolic events)
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with pomalidomide
* Known positive patients for infectious hepatitis, type A, B, C
* Active graft-versus-host disease (GVHD) following allogeneic stem cell transplant for non-AML condition (ex. MDS, MPN, lymphoid malignancy, aplastic anemia) requiring ongoing use of immunosuppressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of pomalidomide, defined as the highest dose at which 0 or 1 dose-limiting toxicities are observed in 6 patients by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (5.0 beginning April 1, 2018) | Up to 21 days
  The proportion of dose-limiting toxicities at each dose level will be reported with exact binomial 95% confidence intervals. Adverse events will be summarized by dose level for all doses. All toxicities by type and grade will be reported.

SECONDARY OUTCOMES:
Proportion of toxicities in the expansion cohort graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (5.0 beginning April 1, 2018) | Up to 2 years
  The proportion of toxicities by type and grade in the expansion cohort will be reported with exact binomial 95% confidence intervals.
Proportion of patients achieving complete remission, complete remission with incomplete count recovery, or partial remission | Up to 2 years
  The proportion of patients achieving each category of response will be reported with 95% exact binomial confidence intervals.
Progression-free survival | Time from start of treatment to time of progression or relapse or death, assessed up to 2 years
  Standard life table methods will be used to analyze progression-free survival. One-year and median progression-free survival with 95% confidence intervals will be reported.
Overall survival | Time of enrollment onto this study to the time of death, assessed up to 2 years
  Standard life table methods will be used to analyze overall survival.

OTHER OUTCOMES:
Change in lymphocyte subpopulations | Baseline to up to 1 year
  Boxplots and line plots will be used to visual trends in the lymphocyte subpopulations. Changes and percentage changes in variables will be summarized. 95% confidence intervals will be obtained by exponentiating the endpoints of confidence intervals for the differences of mean logarithms. A regression model using generalized estimating equations or mixed model used to assess T cell changes. Association of bone marrow and peripheral blood measurements assessed using scatterplots and Spearman's rank correlation coefficients.
Change in levels of antigen-specific CD8+ T cell responses | Baseline to up to 1 year
  McNemar's test will be used to compare proportions with positive tumor specificity before and after pomalidomide treatment. Sensitivity and specificity of induction responses for predicting complete remission status will be estimated.
Presence of minimal residual disease-leukemic stem cells in marrow | Day 14
  Presence or absence of minimal residual disease on day 14 will be correlated with minimal residual disease following induction pomalidomide. McNemar's test will be used to compare proportions. Presence or absence of residual leukemic stem cells immediately following induction will be correlated with progression-free survival using the Kaplan-Meier survival method.
Change in level of cereblon expression in acute myeloid leukemia cells and sorted T cells | Baseline to up to 1 year
  Will examine in relation to clinical parameters as well as T cell reconstitution.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gojo, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina